CLINICAL TRIAL: NCT05854745
Title: Comparison of Virtual Training to In-Person Training of Helping Babies Breathe in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Jimma University (Other); Laerdal Foundation (Other)
Responsible Party: Principal Investigator, Rishi Mediratta, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 62973
Record Dates: First submitted 2023-04-27; First posted 2023-05-11 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Neonatal Death; Birth Asphyxia
Keywords: Helping Babies Breathe (HBB) training
MeSH Terms: conditions — Perinatal Death; Asphyxia Neonatorum

STUDY DESIGN:
Intervention Model Description: The content of each arm of the study is the same and will be taught live by the same HBB instructors; the only difference is the teaching method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual HBB Teaching (Experimental): HBB Virtual Training (Intervention): Participants will receive a blend of virtual training and telesimulation delivered by pediatricians from Ethiopia. The intervention consists of one day of virtual lectures and didactics from the HBB curriculum and skill assessments using neonatal mannequins.
  Interventions: Behavioral: HBB Virtual Training
- In-person HBB Teaching (Active Comparator): Participants will receive in-person HBB instruction by pediatricians from Ethiopia. The control consists of one day of HBB lectures and didactics and skill assessments using neonatal mannequins.
  Interventions: Behavioral: HBB In-person Training

INTERVENTIONS:
Behavioral: HBB Virtual Training — HBB Virtual Training (Intervention): The 2nd edition HBB training course focuses on preparation for birth, routine care for all babies, the Golden Minute, and continued ventilation with normal or slow heart rate. The one-day virtual training will be delivered remotely to participants via Zoom. Facilitators and training materials will be the same in both the control and intervention arms.
  Arms: Virtual HBB Teaching
Behavioral: HBB In-person Training — HBB In-Person Training (Control): The 2nd edition HBB training course focuses on preparation for birth, routine care for all babies, the Golden Minute, and continued ventilation with normal or slow heart rate. The one-day in-person training will be delivered in person. Facilitators and training materials will be the same in both the control and intervention arms.
  Arms: In-person HBB Teaching

SUMMARY:
Helping Babies Breathe (HBB) is a program that teaches providers in low- and middle-income countries about neonatal resuscitation. Historically, HBB training was delivered in person. During the COVID-19 pandemic, many subject matter experts were unable to travel to conduct HBB courses. Innovative methods for teaching HBB are needed to promote the acquisition and retention of resuscitation skills and knowledge.

DETAILED DESCRIPTION:
In this non-inferiority randomized controlled trial, medical students, nursing students, and midwifery students will be randomized to receive either standard in-person HBB training (control) or virtual telesimulation training (intervention). The hypothesis is that virtual delivery is as effective as in-person training of HBB content when teaching neonatal resuscitation skills and knowledge to medical, nursing, and midwifery students.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Year IV through year VI medical students, year II to IV nursing students, year II and III midwifery students at Jimma University in Jimma, Ethiopia.

Exclusion Criteria:

* Minors
* Individuals who are not medical students, nursing students, or midwifery students at Jimma University.
* Individuals who attended a neonatal resuscitation training course in the preceding year.
* Individuals who would be unavailable or unwilling to participate in follow-up study activities throughout the 2-month post-initial training period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Helping Babies Breathe Objective Structured Clinical Exam (OSCE) B | Two months after HBB training (approximately 15 minutes to assess)
  Compare skill retention between the virtual delivery of Helping Babies Breathe (HBB) with the in-person delivery of HBB. This is a standardized evaluation of HBB skills, a score of 17 out of 23 is required to pass. Score range: 0 to 23, higher scores indicate better HBB skills, and a score of 17 or higher is required to pass.

SECONDARY OUTCOMES:
Helping Babies Breathe Objective Structured Clinical Exam (OSCE) B | Immediately after HBB training (approximately 15 minutes to assess)
  Compare skill acquisition between the virtual delivery of Helping Babies Breathe (HBB) with the in-person delivery of HBB. This is a standardized evaluation of HBB skills, a score of 17 out of 23 is required to pass. Score range: 0 to 23, higher scores indicate better HBB skills, and a score of 17 or higher is required to pass.
Helping Babies Breathe Objective Structured Clinical Exam (OSCE) A | Two months after HBB training (approximately 10 minutes to assess)
  Compare skill retention between the virtual delivery of Helping Babies Breathe (HBB) with the in-person delivery of HBB. This is a standardized evaluation of HBB skills, a score of 9 out of 12 is required to pass. Score range: 0 to 12, higher scores indicate better HBB skills, and a score of 9 or higher is required to pass.
Helping Babies Breathe Objective Structured Clinical Exam (OSCE) A | Immediately after HBB training (approximately 10 minutes to assess)
  Compare skill acquisition between the virtual delivery of Helping Babies Breathe (HBB) with the in-person delivery of HBB. This is a standardized evaluation of HBB skills, a score of 9 out of 12 is required to pass. Score range: 0 to 12, higher scores indicate better HBB skills, and a score of 9 or higher is required to pass.
Helping Babies Breathe Bag and Mask Ventilation score | Immediately after HBB training (approximately 10 minutes to assess)
  Compare skill acquisition between virtual delivery of Helping Babies Breathe (HBB) with the in-person delivery of HBB. This is a standardized evaluation of bag and mask ventilation, a score out of 14. Score range: 0 to 14, higher scores indicate better HBB skills, and a score of 14 is required to pass.
Helping Babies Breathe Bag and Mask Ventilation score | Two months after HBB training (approximately 10 minutes to assess)
  Compare skill retention between virtual delivery of Helping Babies Breathe (HBB) with the in-person delivery of HBB. This is a standardized evaluation of bag and mask ventilation, a score out of 14. Score range: 0 to 14, higher scores indicate better HBB skills, and a score of 14 is required to pass.
Helping Babies Breathe Multiple Choice Questionnaire score | Immediately before HBB training (approximately 20 minutes to assess)
  Determine baseline understanding of HBB material for each participant. This exam contains 18 questions pertaining to HBB curriculum. Score range: 0 to 18, higher scores indicate better HBB knowledge, and a score of 15 or higher is required to pass.
Helping Babies Breathe Multiple Choice Questionnaire score | Immediately after HBB training (approximately 20 minutes to assess)
  Determine knowledge acquisition of HBB material for each participant. This exam contains 18 questions pertaining to HBB curriculum. Score range: 0 to 18, higher scores indicate better HBB knowledge, and a score of 15 or higher is required to pass.
Helping Babies Breathe Multiple Choice Questionnaire score | Two months after HBB training (approximately 20 minutes to assess)
  Determine knowledge retention of HBB material for each participant. This exam contains 18 questions pertaining to HBB curriculum. Score range: 0 to 18, higher scores indicate better HBB knowledge, and a score of 15 or higher is required to pass.
NeoNatalie Live Data: Heart rate | Immediately after HBB training (approximately 10 minutes to assess)
  NeoNatalie Live is a mannequin that will provide data on bag-mask ventilation proficiency. During each simulation, the heart rate of the mannequin will be collected per participant.
NeoNatalie Live Data: Ventilation pressure | Immediately after HBB training (approximately 10 minutes to assess)
  NeoNatalie Live is a mannequin that will provide data on bag-mask ventilation proficiency. During each simulation, the ventilation pressure of the mannequin will be collected per participant.
NeoNatalie Live Data: Time to spontaneous breathing | Immediately after HBB training (approximately 10 minutes to assess)
  NeoNatalie Live is a mannequin that will provide data on bag-mask ventilation proficiency. Data about the amount of time it takes to reach a ventilation rate of 40-60 breaths per minute will be collected per participant.
NeoNatalie Live Data: Ventilation attempts | Immediately after HBB training (approximately 10 minutes to assess)
  NeoNatalie Live is a mannequin that will provide data on bag-mask ventilation proficiency. Data about the number of ventilation attempts will be collected per participant.
NeoNatalie Live Data: Heart rate | Two months after HBB training (approximately 10 minutes to assess)
  NeoNatalie Live is a mannequin that will provide data on bag-mask ventilation proficiency. During each simulation, the heart rate of the mannequin will be collected per participant.
NeoNatalie Live Data: Ventilation pressure | Two months after HBB training (approximately 10 minutes to assess)
  NeoNatalie Live is a mannequin that will provide data on bag-mask ventilation proficiency. During each simulation, the ventilation pressure of the mannequin will be collected per participant.
NeoNatalie Live Data: Time to spontaneous breathing | Two months after HBB training (approximately 10 minutes to assess)
  NeoNatalie Live is a mannequin that will provide data on bag-mask ventilation proficiency. Data about the amount of time it takes to reach a ventilation rate of 40-60 breaths per minute will be collected per participant.
NeoNatalie Live Data: Ventilation attempts | Two months after HBB training (approximately 10 minutes to assess)
  NeoNatalie Live is a mannequin that will provide data on bag-mask ventilation proficiency. Data about the number of ventilation attempts will be collected per participant.
Attitude Questionnaire | Immediately before HBB training (approximately 5 minutes to assess)
  5-point Likert scale designed to assess perceived confidence in performing HBB skills.
Attitude Questionnaire | Immediately after HBB training (approximately 5 minutes to assess)
  5-point Likert scale designed to assess perceived confidence in performing HBB skills as well as evaluation satisfaction with the course and its instructors.
Attitude Questionnaire | Two months after HBB training (approximately 5 minutes to assess)
  5-point Likert scale designed to assess sustained perceived confidence in performing HBB skills as well as evaluation satisfaction with the course and its instructors.
Profile of perceived barriers and facilitators | Two months after HBB training (approximately 60 minutes to assess)
  Focus group discussions will be intended to understand differences in perceived barriers/facilitators of training. This will explore confidence in performing HBB techniques and attitudes toward virtual and in-person delivery of content. The objective of the focus groups will be to identify key themes around participants' perspectives of the HBB training to provide context around the outcomes listed above.

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Mediratta, Study Chair — Stanford University
Locations (1):
- Jimma University, Jimma, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data and data dictionary will be available on Dryad within 12 months of publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual de-identified participant data and data dictionary will be available on Dryad within 12 months of publication.
Access Criteria: Data will be shared with researchers upon reasonable request.

REFERENCES:
- [Background] Sobelman C, Richard K, McQuilkin P, Fahey N. Adapting Helping Babies Breathe into a Virtual Curriculum: Methods, Results, and Lessons Learned. Glob Pediatr Health. 2021 May 31;8:2333794X211019698. doi: 10.1177/2333794X211019698. eCollection 2021. PMID 34104697
- [Background] Jones-Bamman C, Niermeyer S, McConnell K, Thomas JF, Olson C. Teaching Helping Babies Breathe via Telehealth: A New Application in Rural Guatemala. Biomed Hub. 2019 Sep 24;4(3):1-6. doi: 10.1159/000502934. eCollection 2019 Sep-Dec. PMID 31993430
- [Derived] Mediratta RP, Clary MK, Liang JW, Daniels K, Muhe LM, Lee HC, Eshetu B, Berhane M. Remote versus in-person pre-service neonatal resuscitation training: A noninferiority randomized controlled trial in Ethiopia. Resuscitation. 2025 Apr;209:110556. doi: 10.1016/j.resuscitation.2025.110556. Epub 2025 Feb 20. PMID 39986344